CLINICAL TRIAL: NCT06356805
Title: Therapeutic Effect of Repetitive Transcranial Magnetic Stimulation on Cognitive and Psychiatric Dysfunction in Patients With Fibromyalgia: A Double Blinded, Randomized Clinical Trial
Brief Title: rTMS Effect on Cognitive and Psychiatric Dysfunction in Patients With Fibromyalgia
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, professor of neurology/Faculty of medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS in Fibromyalgia
Record Dates: First submitted 2024-03-31; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Treatment Resistant Disorders
Keywords: rTMS; FIBROMYALGIA; Hamilton depression and Anxiety scale; MoCa; DLPFC
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Active rTMS of 1 Hz at an intensity of 120% RMT for 60 seconds(20 Trains), with a 45-second gap between trains giving a total of 1,200 pulses/day with the center of coil over rt DLPFC (5cm anterior to hand area). Five sessions/week for 4 consecutive weeks were applied
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): Sham rTMS of 1 Hz at an intensity of 120% RMT for 60 seconds (20 Trains), with a 45-second gap between trains giving a total of 1,200 pulses/day with the coil held perpendicular to the rt DLPFC (5cm anterior to hand area). Five sessions/week for 4 consecutive weeks were applied.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Parallel study: Participants are assigned to one of two groups in parallel for 3 months follow up

SUMMARY:
the aim of this work was to evaluate the effect of low frequency rTMS over the right dorsolateral prefrontal area (DLPFC) on Fibromyalgia patients. Fibromyalgia Impact Questionnaire (FIQ), Hamilton depression and Anxiety scale and different cognitive rating scales were evaluated pre-1 month post sessions and pre -post 3 months later. all eligible patients with fibromyalgia (FM) were randomized to have 20 sessions of active or sham rTMS over right DLPFC. The improvement changes in groups were compared in each rating scale.

DETAILED DESCRIPTION:
The present study was aimed to evaluate the effect of low frequency rTMS over the right dorsolateral prefrontal area (DLPFC) on Fibromyalgia patients. recruitment of the patients were consecutively. Impact Questionnaire (FIQ), psychiatric and cognitive scales were evaluated before rTMS. 42 eligible patients with fibromyalgia (FM) were randomly assigned to one of two groups with equal ratio. each patient received 20 sessions of active or sham rTMS (1 Hz, 120% of resting motor threshold with total 1200 pules /session) over right DLPFC. follow up of each patient was done blindly at , one and 3 months later with the same rating scales (FIQ, Hamilton depression and anxiety Rating Scales (HDRS and HARS), Montreal Cognitive Assessment (MoCA), Rey Auditory Verbal Learning Test (RAVLT), Tower of London test (TOL), the Trail Making and Digit Span Tests). comparison between the changes in different rating scales were done at 1- and 3-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of fibromyalgia was made according to American College of Rheumatology criteria with age at and older than 18 years

Exclusion Criteria:

Inflammatory rheumatic disease, auto immune disease, or other painful disorders. Any uncontrolled clinical disease (such as thyroid, cardiovascular, pulmonary, hematological, or renal disease) that affects cognition. Pregnancy, lactation. patients have one of Contra-indications for rTMS (a history of seizures, brain trauma, brain surgery or intracranial hypertension, a pacemaker, or other metallic implants), Past history of other neurological disorders (neurodegenerative diseases, dementia), or primary psychiatric disorders (psychosis, or major depression (17-item Hamilton Depression Rating Scale > 23), or drug treatments that affect cognition. Inability to cooperate with the questionnaire survey or the patient refuses to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
1- Assessment of Fibromyalgia Impact Questionnaire (FIQ) | 3 months
  Assessment of the changes (pre-post one month and pre- post three months later) in Fibromyalgia Impact Questionnaire FIQ. It is a brief 10-item self-administered instrument that takes approximately 5 minutes to complete. It has been designed to measure physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and wellbeing. The average FM patient scores about 50, severely afflicted patients are usually 70 plus.

SECONDARY OUTCOMES:
1-Assessment of Hamilton depression (HDRS) and Hamilton Anxiety scales (HARS) (pre- post sessions and pre post three months) | 3 months follow up
  Assessment of the changes (pre-post one month and pre- post three months later) of HDRS and HARS in Fibromyalgia patients. It contains 17 items (HDRS) pertaining to symptoms of depression experienced over the past week. The HARS consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety and somatic anxiety (physical complaints related to anxiety).
Assessment of different cognitive rating scales (Montreal cognitive Assessment scale (MoCa), and Rey Auditory Verbal Learning Test [RAVLT], | 3 months follow up
  Assessment the changes of different cognitive rating scales (pre-post sessions and pre- post three months later) in fibromyalgia patients.
  MoCa takes 10 to 12 minutes to complete. It based on 11 questions that evaluate seven domains of cognitive function. The MoCa has a maximum score of 30, and anything below 24 is a sign of cognitive impairment.
  RAVLT: it consists of five presentations of a 15-word list are given, each followed by attempted recall. This is followed by a second 15-word interference list (list B), followed by recall of list A. The number of correct words summed for the Total Recall score (range = 0-75). The Delayed Recall score is the number of correct words recalled after a 30-min delay (range = 0-15).

CONTACTS AND LOCATIONS:
Overall Officials: Eman Khedr, professor, Principal Investigator — Assiut University
Locations (1):
- Eman Khedr, Asyut, Egypt